CLINICAL TRIAL: NCT03269162
Title: The Prognosis Study of Postoperative Non-small-cell Lung Cancer Patients Treated Precisely With the Integrated Traditional Chinese and Western Medicine Based on CTC Detection
Brief Title: Postoperative NSCLC Treated With Integrated Medicine Base on Circulating Tumor Cell Detection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: lihegen (Other)
Responsible Party: Sponsor-Investigator, lihegen, Director of Oncology Department Longhua Hospital, Shanghai University of Traditional Chinese Medicine
Organization: Shanghai University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHDC12016114
Record Dates: First submitted 2017-08-18; First posted 2017-08-31 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: NSCLC
MeSH Terms: interventions — Docetaxel; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jinfukang + Chemotherapy Group (Experimental)
  Interventions: Drug: Jinfukang Koufuye; Drug: Docetaxel; Drug: Pemetrexed; Drug: Cisplatin
- Chemotherapy Group (Placebo Comparator)
  Interventions: Drug: Docetaxel; Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: Jinfukang Koufuye — 30ml per time, tid, po (d6-21, q21)
  Arms: Jinfukang + Chemotherapy Group
Drug: Docetaxel — 75mg/m2,ivgtt 30mins, d1
Drug: Pemetrexed — 500mg/m2, ivgtt 30mins, d1
Drug: Cisplatin — 75mg/m2, ivgtt >2h, d1

SUMMARY:
Objective: To study the effect of Jinfukang Koufuye combined with chemotherapy on preventing relapse and metastasis of early postoperative NSCLC patients. Method: In this multicenter、prospective、randomized controlled clinical trial, 144 NSCLC patients with complete resection、stage Ib-IIb were randomly divided into Jinfukang Koufuye combined with chemotherapy group (treatment group, N=72) and chemotherapy only group (controlled group, N=72). Peripheral blood CTCs and immune cells were detect on five different time points: after operation、4 chemotherapy cycles were over、12 months after operation、18 months after operation、and 24 months after operation. To evaluate the effect of Jinfukang Koufuye combined with chemotherapy on the level of peripheral blood CTCs、DFS、immune function、quality of life of postoperative patients; and decreasing the side effect of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Pathology-confirmed diagnosis of primary NSCLC with complete resection, and stage IB-IIB
2. Accept chemotherapy for the first time 6 weeks after operation
3. Age of 18-75 years old
4. Eastern Cooperative Oncology Group-PS≤2
5. N>1.5×109/L、PLT> 100 × 109/L、Hb>100g/dL、Liver and kidney function is normal or elevated ≤ 1.5 times
6. Voluntary participation in the prospective study with signed informed consent

Exclusion Criteria:

1. No pathology-confirmed diagnosis patients
2. Patients with overall survival time<6 months
3. Patients with Serious diseases like heart、liver、kidney and hematopoietic system at the same time
4. Pregnant or breast feeding patients
5. Patients with uncontrollable mentally disease
6. Patients with diabetes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2016-09-30 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival Rate | 2 years
  From the very beginning of the randomization to the end point when disease relapse or death because of any reason

CONTACTS AND LOCATIONS:
Overall Officials: Hegen Li, Principal Investigator — Longhua Hospital